CLINICAL TRIAL: NCT01075308
Title: A Phase II Study of SB939 in Patients With Recurrent or Metastatic Castration Resistant Prostate Cancer
Brief Title: SB939 in Treating Patients With Recurrent or Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: S*BIO (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I195; CAN-NCIC-IND195 (Registry Identifier: NCI US PDQ); CDR0000666241 (Other: PDQ)
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Prostate Cancer
Keywords: hormone-resistant prostate cancer; recurrent prostate cancer; stage IV prostate cancer; stage III prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — SB939 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SB939 (Experimental): SB939 given orally every other day 3 times a week (i.e. Monday /Wednesday /Friday, or Tuesday /Thursday / Saturday) for 3 consecutive weeks followed by one week off-dosing. A treatment cycle is 4 weeks (28 days).
  Interventions: Drug: HDAC inhibitor SB939

INTERVENTIONS:
Drug: HDAC inhibitor SB939 — SB939 given orally every other day 3 times a week (i.e. Monday /Wednesday /Friday, or Tuesday /Thursday / Saturday) for 3 consecutive weeks followed by one week off-dosing. A treatment cycle is 4 weeks (28 days).

SUMMARY:
RATIONALE: SB939 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well SB939 works in treating patients with recurrent or metastatic prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the efficacy, as measured by PSA response and progression-free survival, of HDAC inhibitor SB939 in patients with recurrent or metastatic castration-resistant prostate cancer.

Secondary

* To determine the objective response and response duration in patients with measurable disease at baseline.
* To determine the tolerability and toxicity of this drug in these patients.
* To determine the number of circulating tumor cells at baseline and after 6 weeks (and 12 weeks if patient is still on study treatment).
* To explore potential molecular factors predictive of response by assessment of archival prostate tumor tissue.
* To explore ERG and PTEN expression on circulating tumor cells as a potential prognostic and predictive marker for response to this drug.
* To determine time to PSA and time to objective progression in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral HDAC Inhibitor SB939 once daily on days 1, 3, 5, 8, 10, 12, 15, 17, and 19. Treatment repeats every 4 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for correlative studies. Blood samples and Archival tumor tissue are analyzed for TMPRSS2-ERG fusion and PTEN deletion status by FISH; TMPRSS2-ERG fusion by RT-PCR; and for the number of circulating tumor cells.

After completion of study therapy, patients are followed up at 4 weeks and then every 3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate
* Presence of clinically and/or radiologically documented disease (target or non-target)
* Metastatic or locally recurrent disease for which no curative therapy exists AND for which systemic chemotherapy is indicated due to progression, meeting the following criteria:

  * At least two rises in PSA over a reference value OR the development of new metastatic lesions with a stable or rising PSA

    * First rising PSA must be taken at least 1 week after the reference value
    * Third or subsequent PSA must show further increase confirming progression within 2 weeks prior to study enrollment
    * PSA progression must be documented after discontinuation of peripheral antiandrogens (4 weeks for flutamide and 6 weeks for bicalutamide/nilutamide) for patients with documented evidence of progression while receiving peripheral antiandrogens
* Medically or surgically castrated by androgen ablation

  * Castrate level of testosterone (< 1.7 nmol/L) must be present for patients undergoing medical androgen ablation
* Received prior hormone therapy

  * Must have hormone-refractory disease
  * Therapy with luteinizing hormone-releasing hormone (LHRH) agonist must continue for patients already receiving this treatment at the time of enrollment
  * Patients who discontinued LHRH agonist must restart therapy (if not surgically castrated) and the castrate level of testosterone must be present
* PSA ≥ 5 ng/mL
* Primary or metastatic tumor tissue available
* No documented CNS metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 12 weeks
* Absolute granulocyte count ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin normal
* Serum creatinine normal
* Potassium normal
* Calcium normal
* Fertile patients must use effective contraception
* QTc ≤ 450 msec
* LVEF ≥ 50% by Echo or MUGA scan
* Troponin I or T ≤ ULN
* Able to take oral medication
* No preexisting uncontrolled cardiac condition
* No prior myocardial infarction
* No history of other malignancies, except adequately treated nonmelanoma skin cancer or other solid tumors curatively treated with no evidence of disease for ≥ 5 years
* No gastrointestinal abnormalities (e.g., bowel obstruction or previous gastric resection) that would lead to inadequate absorption of HDAC Inhibitor SB939
* No known HIV positivity or hepatitis B or C infections
* No chronic medical condition or comorbidity that may increase the risks associated with study participation/study drug administration or may interfere with the interpretation of study results, including any of the following:

  * Pulmonary disease
  * Active infection
  * Psychiatric condition
  * Laboratory abnormality

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior antiandrogens (6 weeks for bicalutamide)
* At least 4 weeks since prior external-beam radiotherapy

  * Exceptions may be made for low-dose, non-myelosuppressive radiotherapy
* At least 28 days since other prior investigational therapy or anticancer therapy
* At least 14 days since prior major surgery and wound healing has occurred
* No more than 1 prior chemotherapy regimen allowed and recovered from significant toxicity
* No prior strontium
* No prior HDAC inhibitors
* No current agents (dysrhythmic drugs) with a known risk of Torsades de Pointes
* No other concurrent cytotoxic therapy or radiotherapy
* No other concurrent investigational therapy

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-06-28 (Actual); Primary Completion 2015-01-05 (Actual); Study Completion 2015-02-13 (Actual)

PRIMARY OUTCOMES:
PSA response | each cycle
  Each patient will have PSA response calculated. Required at the end of every cycle.
Progression-free survival | end of study
  Used as an indicator of efficacy, patients with PSA response will have length of progression free survival calculated.

SECONDARY OUTCOMES:
Objective response rate | every other cycle
  Patients with measurable disease will have objective response evaluated.
Duration of response | every other cycle
  Patients with objective response will have duration of response calculated as will be followed until progression/relapse
Safety | each cycle
  Toxicity and tolerability will be evaluated
Change in circulating tumor cells during study compared to baseline | each cycle
  Patients will have on study samples compared to baseline to look for chance in number of CTC.
Comparison of TMPRSS2-ERG fusion and PTEN deletion in circulating tumor cells | each cycle
  samples will be taken and analyzed each cycle with a comparison made at end of study.
Comparison of two systems for counting circulating tumor cells | end of study
  Two different systems will be used to count CTC. Results will be compared at the end of the study for accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Kim N. Chi, MD, Study Chair — British Columbia Cancer Agency; Bernhard Eigl, MD, FRCPC, Study Chair — Tom Baker Cancer Centre - Calgary
Locations (7):
- Canada (7):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - London Regional Cancer Program, London, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eigl BJ, North S, Murray N, Heng DYC, Winquist E, Powers J, Walsh WR, Eisenhauer E, Squire J, Cox M, Chi KN. A Phase II Study of SB939 in Patients with Recurrent or Metastatic Castration Resistant Prostate Cancer (CRPC). AACR Mol Cancer Tehr 10[11 Suppl; abstr A211]. 2011
- [Result] Eigl BJ, North S, Murray N, Heng DYC, Winquist E, Powers J, Walsh WR, Eisenhauer E, Squire J, Cox M, Chi KN. A Phase II Study of SB939 in Patients with Recurrent or Metastatic Castration Resistant Prostate Cancer (CRPC). Canadian Cacner Research Conference. 2011.
- [Result] Eigl BJ, North S, Winquist E, Finch D, Wood L, Sridhar SS, Powers J, Good J, Sharma M, Squire JA, Bazov J, Jamaspishvili T, Cox ME, Bradbury PA, Eisenhauer EA, Chi KN. A phase II study of the HDAC inhibitor SB939 in patients with castration resistant prostate cancer: NCIC clinical trials group study IND195. Invest New Drugs. 2015 Aug;33(4):969-76. doi: 10.1007/s10637-015-0252-4. Epub 2015 May 19. PMID 25983041